CLINICAL TRIAL: NCT01369303
Title: Pharmacokinetic and Pharmacodynamic Study of Tenofovir 1% Gel Using the Bat 24 Regimen Versus Daily and Pericoital Dosing
Brief Title: Pharmacokinetic and Pharmacodynamic Study of Tenofovir 1% Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A10-113
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Prevention
Keywords: HIV
MeSH Terms: interventions — Tenofovir; Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Daily dosing (Experimental): Tenofovir 1% gel will be inserted each day or evening at about the same time with the last study-sex 12 hours after the final dose
  Interventions: Drug: Tenofovir 1% vaginal gel
- BAT24 dosing (Experimental): Tenofovir 1% gel will be inserted 1 hour before and 1 hour after sex
  Interventions: Drug: Tenofovir 1% vaginal gel
- Pericoital dosing (Experimental): Tenofovir 1% gel will be inserted either 1 hour before sex OR 1 hour after sex
  Interventions: Drug: Tenofovir 1% vaginal gel

INTERVENTIONS:
Drug: Tenofovir 1% vaginal gel — Tenofovir 1% gel is supplied as a clear, transparent, viscous gel packaged in pre-filled single use applicators. Each applicator contains 4.0 mL of tenofovir gel (equal to 4.4 gm) at a concentration of 1% (weight for weight) formulated in purified water with edetate disodium, citric acid, glycerin, methylparaben, propylparaben and hydroxyethylcellulose, and is pH adjusted to 4-5.

SUMMARY:
The purpose of the study is to obtain data on the pharmacokinetics (PK) and pharmacodynamics (PD) and immune system effect of the BAT24 dosing regimen versus daily and pericoital dosing regimens with vaginal use of tenofovir 1% gel after a single sex act and after multiple sex acts.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years, inclusive;
* General good health (by volunteer history and per investigator discretion) without any clinically significant systemic disease (including, but not limited to, significant liver disease/hepatitis, gastrointestinal disease, kidney disease, thyroid disease, osteoporosis or bone disease, and type 2 diabetes);
* Currently having regular menstrual cycles, if not on hormonal (including continuous) contraception, by volunteer report and per investigator discretion;
* History of Pap smears and follow-up consistent with American Congress of Obstetricians and Gynecologist (ACOG) practice guideline #109 (see study manual) or willing to undergo a Pap smear at Visit 1. (Note: See study manual for clarification of eligibility criteria specific to Pap smear results.)
* Willing to abstain from the use of any vaginal product other than the study gel including spermicides, lubricants, vaginal hygiene products, contraceptive intravaginal ring, diaphragms, and cervical caps (non-hormonal IUC if used as her method of contraception, is allowed) for the duration of the study;
* In a monogamous relationship for at least the last four months with a male partner, at least 18 years old with no known risks for STIs, and not known to be HIV positive, who is willing and able to comply with the study requirements, and with whom condoms are not typically used;
* Protected from pregnancy by sterilization of either partner, use of combination oral contraceptives or patch for at least two cycles, or non-hormonal intrauterine contraception throughout the study. Continuous oral contraceptives are allowable if the patient is at low risk for breakthrough bleeding;
* Vaginal and cervical anatomy that, in the opinion of the investigator, lends itself to easy genital tract sample collection;
* Negative urine pregnancy test; and
* Willing to give voluntary consent, sign an informed consent form and comply with study procedures as required by the protocol.

Exclusion Criteria:

* History of hysterectomy;
* Currently pregnant or within two calendar months from the last pregnancy outcome. Note: If recently pregnant must have had at least two spontaneous menses since pregnancy outcome;
* Use of Depo-Provera in the last 120 days;
* Currently breastfeeding or having breastfed an infant in the last two months, or planning to breastfeed during the course of the study;
* History of sensitivity/allergy to any component of the study product, topical anesthetic, or allergy to both silver nitrate and Monsel's solution;
* In the last six months, diagnosed with or treated for any STI or pelvic inflammatory disease. Note: Women with a history of genital herpes or condylomata who have been asymptomatic for at least six months may be considered for eligibility;
* Symptomatic vulvovaginal candidiasis, Nugent score greater than equal to 7 at screening or symptomatic bacterial vaginosis (BV) at Visit 2, or symptomatic urinary tract infection (UTI);
* Positive test for Trichomonas vaginalis, Neisseria gonorrhea or Chlamydia trachomatis;
* Deep epithelial genital findings such as abrasions, ulcerations, and lacerations, or vesicles suspicious for a sexually transmitted infection;
* Positive test for HIV;
* Positive test for Hepatitis B surface antigen (HBsAg);
* Known bleeding disorder that could lead to prolonged or continuous bleeding with biopsy;
* Chronic or acute vulvar or vaginal symptoms (pain, irritation, spotting, etc.);
* Known current drug or alcohol abuse which could impact study compliance;
* Grade 1 or higher laboratory abnormality, per the August 2009 update of the DAIDS Table for Grading the Severity of Adverse Events;
* Systemic use in the last two weeks or anticipated use during the study of drugs on a daily basis that may reduce renal function (e.g., ibuprofen) or liver function (e.g., Tylenol®), or that may affect anti-HSV activity (e.g., acyclovir or valacyclovir) of any of the following: corticosteroids, antibiotics, antifungals, antivirals (e.g. acyclovir or valacylovir) or antiretrovirals (e.g. Viread®). Note: Participants should avoid nonsteroidal anti-inflammatory drugs (NSAIDs) except for treatment of dysmenorrhea during menses. Participants may use Tylenol® on an as-needed but not daily basis during the study
* Participation in any other investigational trial (device, drug, or vaginal trial)within the last 30 days for this study or planned participation in any other investigational trial during the study;
* History of gynecological procedures (including genital piercing) on the external genitalia, vagina or cervix within the last 14 days; and
* Abnormal finding on laboratory or physical examination or a social or medical condition which, in the opinion of the investigator, would make participation in the study unsafe or would complicate interpretation of data.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 194 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
TFV concentrations in blood plasma, aspirate and tissue and TFV-DP concentrations in PBMCs, endocervical cells and tissue to evaluate if a single precoital or postcoital dose provides concentrations similar to BAT24 after a single sex act. | Assigned time-point after a single act of study-related sex
  Each participant will be randomized to one of nine groups: (dosing regimen: BAT24, precoital or postcoital) x (sample collection time-point: 4, 12 or 72 hours after the single act of study-related sex). Approximately 30 women will be assigned to each dosing regimen.
TFV concentrations in blood plasma, aspirate and tissue and TFV-DP concentrations in PBMCs, endocervical cells and tissue to evaluate if daily or intermittent pericoital dosing provides concentrations similar to BAT24 after two weeks of twice weekly sex | Assigned time-point after the last act of study-related sex
  Participants will be randomized to 1 of 12 groups: (dosing regimen: BAT24, precoital, postcoital or daily) x (sample collection time-point: 4, 12 or 72 hrs after the last act of study-related sex). 30 women will be assigned to each the BAT24 and daily dosing regimens; 15 will be assigned to each the pre- and postcoital dosing regimens. Those assigned to the BAT24 or a pericoital regimen will have study-related sex twice weekly for 2 weeks. Those assigned to the daily regimen will use the gel at about the same time each day for 2 weeks and to have sex at least twice each week.

SECONDARY OUTCOMES:
Characterize anti-HIV and anti-HSV activity of cervicovaginal lavages (CVLs) at baseline and after a single sex act using BAT24 and a single precoital or postcoital dose of TFV gel | Assigned time-point after a single act of study-related sex
Anti-HIV and anti-HSV activity of CVLs after two weeks of twice weekly sex using BAT24, daily and pericoital dosing of TFV gel | Assigned time-point after the last act of study-related sex
Compare genitourinary adverse events (AEs) after administration of TFV gel | Assigned time-point after study-related sex (single act and two weeks of twice weekly study-related sex)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Schwartz, M.D., Study Director — CONRAD
Locations (5):
- United States (4):
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Advances in Health, Inc., Houston, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia
- Profamilia, Santo Domingo, Dominican Republic, Dominican Republic